CLINICAL TRIAL: NCT06271629
Title: Impact of Quality of Life in the Patients With Sleep Disturbance From Low Anterior Resection Syndrome in Advanced Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2204-042-1314
Record Dates: First submitted 2024-02-04; First posted 2024-02-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Rectal Cancer; Low Anterior Resection Syndrome; Insomnia
Keywords: low anterior resection syndrome; insomnia
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Insomnia Severity index Grade 0&1: administered the Insomnia Severity Index (Korean validated version) to patients with Low Anterior Resection Syndrome (LARS) and divided them into two groups based on the severity grade.
  Interventions: Diagnostic Test: Insomnia severity index
- Insomnia Severity index Grade 2&3: administered the Insomnia Severity Index (Korean validated version) to patients with Low Anterior Resection Syndrome (LARS) and divided them into two groups based on the severity grade.
  Interventions: Diagnostic Test: Insomnia severity index

INTERVENTIONS:
Diagnostic Test: Insomnia severity index — The ISI score is a self-report questionnaire consisting of 7 items designed to assess the nature, severity, and impact of insomnia.(16) The typical recall period for respondents is the "last month." The evaluated dimensions include the severity of sleep onset, sleep maintenance, and early morning awakening problems, as well as sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and the distress caused by the sleep difficulties.

SUMMARY:
The preservation surgery of the anal sphincter has become a standard procedure for the treatment of rectal cancer and is now possible even when the tumor is close to the anus, thanks to the advancement of surgical techniques. This procedure allows patients to avoid a permanent artificial anus and enables them to evacuate through the anus, maintaining the continuity of the intestine, making it a highly preferred surgical option. Additionally, advancements in tumor treatments have led to improved long-term survival rates.

However, this anal sphincter preservation surgery inevitably can cause functional abnormalities in the rectum, and around 90% of patients experience changes in bowel habits after surgery. The characteristic symptoms occurring after rectal cancer surgery, such as diarrhea, urgency of bowel movements, frequent bowel movements, and fecal incontinence, are referred to as Anterior Resection Syndrome (ARS). Particularly, symptoms following low anterior resection surgery for lower rectal cancer are termed Low Anterior Resection Syndrome (LARS). These symptoms are most severe immediately after surgery, persisting up to 1-2 years, with some improvement over time. However, in many patients, LARS can remain a lifelong challenge, significantly impacting their quality of life. Currently, there is no definitive method to treat LARS, and symptom management is achieved through empirical treatment methods or medications.

Many patients with LARS experience these symptoms predominantly at night, and it is presumed that their sleep quality is severely compromised, significantly affecting their overall quality of life. However, there is a lack of research on the prevalence of such patients and the appropriate treatments for them.

DETAILED DESCRIPTION:
1. administer the Low Anterior Resection Syndrome (LARS) questionnaire to patients who underwent low anterior resection surgery for progressive rectal cancer and completed anticancer treatment, with a time lapse of approximately 1 month to 5 years.
2. investigate the use of medication or conservative treatment for managing symptoms of Low Anterior Resection Syndrome.
3. assess whether the symptoms captured in the Low Anterior Resection Syndrome questionnaire primarily occur during the day or night by surveying each of the 5 items in the questionnaire. We determine the overall symptom score by adding up the scores for daytime and nighttime symptoms, selecting the higher score.
4. conduct a survey on the quality of sleep.
5. conduct a survey on the quality of life. compiled the results of the questionnaires and analyze the correlations among them.

ELIGIBILITY:
Inclusion Criteria:

* undergone low anterior resection for progressive rectal cancer
* undergone bowel continence restoration surgery and are between 1 month and 5 years postoperative
* ability to comprehend and participate in the clinical trial

Exclusion Criteria:

* A history of previous surgery for colorectal cancer
* Recurrent colorectal cancer
* Concomitant metastatic colorectal cancer
* Requiring permanent colostomy
* Underlying conditions not controlled by medical treatment
* Inflammatory bowel disease
* Chronic constipation or diarrhea not controlled by medication before surgery
* Preoperative symptoms of fecal incontinence
* Preoperative symptoms of bowel leakage
* Allergies to the investigational drug
* Deemed unsuitable for participation in the clinical trial by the principal investigator and study staff

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone low anterior resection surgery following progressive rectal cancer without permanent stoma
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Impairment in the quality of sleep and quality of life in patients with Low Anterior Resection Syndrome (LARS). | 1 Month
  Insomnia Severity Index Score : Sum of Insomnia Severity Index score

SECONDARY OUTCOMES:
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 1 Month
  Symptoms & quality of life evaluation in LARS patients
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-CR29) | 1 Month
  Symptoms & quality of life evaluation in LARS patients

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No